CLINICAL TRIAL: NCT03082326
Title: The Critical Care Ultrasound Based Characteristic of Hemodynamic and Lung Pathology in Early Stage of Shock in ICU: The Epidemic and Prognostic Value
Brief Title: The CCUS Based Characteristic of Hemodynamic and Lung Pathology in Early Stage of Shock in ICU: The Epidemic and Prognostic Value
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, tongjuan ZOU, Doctor, West China Hospital
Other Study IDs: West China H
Record Dates: First submitted 2017-03-03; First posted 2017-03-17 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-03

CONDITIONS: Shock
Keywords: shock; critical care ultrasound; hemodynamics; lung pathology; epidemic; prognosis
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Shock is a common condition in critical care unit (ICU). It is extremely important that the patient accepts early goal-directed therapy (EGDT) treatment in the early stage of shock. However, several studies failed to demonstrate that the well used variables such as CVP and others could direct to a better treatment. In recent years, critical care ultrasound (CCUS) has been respected as a reliable noninvasive tool and widely used in ICU practice. With CCUS the investigators can accurately acquired the detailed information of the characteristic of the hemodynamics and lung pathology (the systole and diastole function, volume status, valve insufficiency, lung, edema, consolidation, and pleural effusion, etc.). To the investigators knowledge, there is no study investigating the epidemic of such ultrasonic variables and its value to predict to outcome. The aim of this study is to investigate the epidemic and the prognostic value of CCUS Based Characteristic of Hemodynamic and Lung pathology in Early Stage of Shock in patients admitted in ICU.

DETAILED DESCRIPTION:
Adult patients who admitted to the intensive care unit of West China hospital of sichuan university with shock from April 2016 to April 2017 enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. SBP<90 mm Hg or MAP <70 mm Hg or SBP decrease >40mmHg or need vasoactive drugs;
2. Skin that is cold and clammy, capillary refill time >4.5s, urine output of <0.5ml/Kg.hr and lactate>2mmol/L;
3. SHOCK presented within 6 hr.

Exclusion Criteria:

1. <18 years old;
2. Pregnancy;
3. Patient or family member refuse to be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Shock patients with 6 hours admitted in ICU in west china hospital of sichuan university.
Sampling Method: Non-Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2016-04-05; Primary Completion 2017-06-06 (Actual); Study Completion 2017-06-06 (Actual)

PRIMARY OUTCOMES:
all cause mortality | 28 days

SECONDARY OUTCOMES:
length of mechanical ventilation | through study completion, an average of 28 days
ICU length of stay | through study completion, an average of 28 days
hospital length of stay | through study completion, an average of 28 days

CONTACTS AND LOCATIONS:
Overall Officials: yan kang, doctor, Study Chair — West China Hospital
Locations (1):
- West China Hospital,Sichuan University, Chengde, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rivers E, Nguyen B, Havstad S, Ressler J, Muzzin A, Knoblich B, Peterson E, Tomlanovich M; Early Goal-Directed Therapy Collaborative Group. Early goal-directed therapy in the treatment of severe sepsis and septic shock. N Engl J Med. 2001 Nov 8;345(19):1368-77. doi: 10.1056/NEJMoa010307. PMID 11794169
- [Result] Vincent JL, De Backer D. Circulatory shock. N Engl J Med. 2014 Feb 6;370(6):583. doi: 10.1056/NEJMc1314999. No abstract available. PMID 24499231
- [Result] Seif D, Perera P, Mailhot T, Riley D, Mandavia D. Bedside ultrasound in resuscitation and the rapid ultrasound in shock protocol. Crit Care Res Pract. 2012;2012:503254. doi: 10.1155/2012/503254. Epub 2012 Oct 24. PMID 23133747
- [Result] Levitov A, Frankel HL, Blaivas M, Kirkpatrick AW, Su E, Evans D, Summerfield DT, Slonim A, Breitkreutz R, Price S, McLaughlin M, Marik PE, Elbarbary M. Guidelines for the Appropriate Use of Bedside General and Cardiac Ultrasonography in the Evaluation of Critically Ill Patients-Part II: Cardiac Ultrasonography. Crit Care Med. 2016 Jun;44(6):1206-27. doi: 10.1097/CCM.0000000000001847. PMID 27182849
- [Result] Guerin L, Vieillard-Baron A. The Use of Ultrasound in Caring for Patients with Sepsis. Clin Chest Med. 2016 Jun;37(2):299-307. doi: 10.1016/j.ccm.2016.01.005. Epub 2016 Mar 3. PMID 27229646
- [Result] Wang H, Cui N, Su L, Long Y, Wang X, Zhou X, Chai W, Liu D. Prognostic value of extravascular lung water and its potential role in guiding fluid therapy in septic shock after initial resuscitation. J Crit Care. 2016 Jun;33:106-13. doi: 10.1016/j.jcrc.2016.02.011. Epub 2016 Feb 24. PMID 27021852
- [Derived] Zhou R, Zou T, Yin W, Wang X, Kang Y; Chinese Critical Ultrasound Study Group (CCUSG). Functional mitral regurgitation combined with increased early diastolic transmitral velocity to early mitral annulus diastolic velocity ratio is associated with a poor prognosis in patients with shock. Chin Med J (Engl). 2021 Sep 15;134(19):2299-2305. doi: 10.1097/CM9.0000000000001756. PMID 34629416
- [Derived] Zou T, Yin W, Li Y, Deng L, Zhou R, Wang X, Chao Y, Zhang L, Kang Y; Chinese Critical Ultrasound Study Group (CCUSG). Hemodynamics in Shock Patients Assessed by Critical Care Ultrasound and Its Relationship to Outcome: A Prospective Study. Biomed Res Int. 2020 Sep 15;2020:5175393. doi: 10.1155/2020/5175393. eCollection 2020. PMID 33015171